CLINICAL TRIAL: NCT03978884
Title: An Open Label, Single Arm Prospective Study to Evaluate Efficacy and Safety of Losartan Based Therapy Reslio® (Losartan) and Resilo-h® (Losartan+Hydrochlorthiazide) in Diabetic and Uncontrolled Hypertensive Patients
Brief Title: Phase 4 Study of the Efficacy of Losartan Based Therapy in Hypertensives With and Without Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to effective arrange trial logistics
Sponsor: The University of The West Indies (Other)
Collaborators: Caribbean College of Family Physicians (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECP231516
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Losartan; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild Hypertensive (Experimental): Mild Hypertensive with systolic BP >=140 mmHg but less than 160 mmHg at baseline with diastolic >=90 but <100 mmHg
  Interventions: Drug: Losartan 50Mg Tab; Drug: Losartan/Hydrochlorothiazide 100 Mg-25 Mg ORAL TABLET
- Mild Hypertensive with Diabetes (Experimental): Mild Hypertensive with systolic BP >=140 mmHg but less than 160 mmHg at baseline with diastolic >=90 but <100 mmHg and diabetes.
  Interventions: Drug: Losartan/Hydrochlorothiazide 50 Mg-12.5 Mg ORAL TABLET; Drug: Losartan/Hydrochlorothiazide 100 Mg-25 Mg ORAL TABLET
- Severe Hypertension (Experimental): Severe Hypertensive with systolic BP >=160 mmHg at baseline or with diastolic >=100 mmHg
  Interventions: Drug: Losartan/Hydrochlorothiazide 100 Mg-25 Mg ORAL TABLET; Drug: Amlodipine 5mg
- Severe Hypertension with Diabetes (Experimental): Severe Hypertensive with systolic BP >=160 mmHg at baseline or with diastolic >=100 mmHg with diabetes
  Interventions: Drug: Losartan/Hydrochlorothiazide 100 Mg-25 Mg ORAL TABLET; Drug: Amlodipine 5mg

INTERVENTIONS:
Drug: Losartan 50Mg Tab — Take 1 tab daily
  Arms: Mild Hypertensive
Drug: Losartan/Hydrochlorothiazide 50 Mg-12.5 Mg ORAL TABLET — Take 1 tab daily
  Arms: Mild Hypertensive with Diabetes
Drug: Losartan/Hydrochlorothiazide 100 Mg-25 Mg ORAL TABLET — Take 1 tab daily
Drug: Amlodipine 5mg — Take 1 tablet daily
  Arms: Severe Hypertension; Severe Hypertension with Diabetes

SUMMARY:
To study antihypertensive efficacy of 12 weeks of Losartan based therapy Resilo (Losartan) and Resilo-H (Losartan+ Hydrochlorothiazide) in uncontrolled hypertensive and diabetic hypertensive patients.

DETAILED DESCRIPTION:
200 hundred Subjects will be treated with a dose escalation regimen to achieve a target blood pressure. Subjects with mild hypertension at baseline will be started with losartan 50 mgs and those with severe hypertension will be started with losartan H 100/25. After 6 weeks they will titrated if goal blood pressure not achieved. For Mild hypertensive group this will be with losartan H 100/25 and for severe hypertensive group this will by addition of amlodipine 5 mg to regime. Subjects with mild hypertension and diabetes at baseline will be started with losartan H 50/12.5 mg and those with severe hypertension with diabetes will be started with losartan H 100/25. After 6 weeks they will be titrated if goal blood pressure not achieved. For Mild hypertensive-diabetic group this will be with Resilo H 100/25 and for severe hypertensive group this will by addition of amlodipine 5 mg to regime.

Target Blood Pressure is systolic < 140 mmhg and diastolic < 90 mmHg if age < 60 years and systolic < 150 mmHg and diastolic < 90 mmHg if age >60 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign Informed Consent Form.
* Patients of either sex above 18 years of age.
* Patients not previously diagnosed with hypertension and with sitting blood pressure > 140/90 mmHg on two readings 15 minutes apart.
* Newly diagnosed hypertensive patients.
* Hypertensive patients on other antihypertensive therapies but not at goal
* Diabetes defined as patient on insulin therapy or oral diabetic therapy or fasting blood glucose on screening > 7 mmol/L

Exclusion Criteria:

* Patients with history of allergic reaction to any angiotensin II antagonist or a thiazide diuretic
* Patients with history suggestive secondary hypertension
* Patients who have taken Resilo or Resilo-H or other losartan based treatment in past three months of study inclusion.
* Patients with chronic renal failure or who on screening has serum creatinine >150 µmol/L
* Patients who is participating concurrently in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects achieving Target Blood Pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Reid, Principal Investigator — University of the West Indies
Locations (1):
- Tropical Metabolism Research Unit, Kingston, Other, Jamaica

IPD SHARING:
Plan to Share IPD: No